CLINICAL TRIAL: NCT03605355
Title: Feasibility Study on the Medical and Economic Consequences of an Ambulatory Transient Ischemic Attack and Minor Stroke Management
Brief Title: Feasibility Study on the Medical and Economic Consequences of Outpatient Management of TIAs and Minor Strokes
Acronym: MEDECO-AIT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0349; 2018-A01444-51 (Other: ID-RCB)
Record Dates: First submitted 2018-07-19; First posted 2018-07-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Transient Ischemic Attack
Keywords: minor stroke; cost-effectiveness; feasibility; day clinic
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effectiveness of outpatient management of minor TIAs and strokes in the context of a dedicated outpatient pathway with specialized care has been demonstrated and has resulted in an 80% decrease in stroke in the year followed the AIT (EXPRESS and SOS-TIA studies) At the same time, few studies have been conducted on their economic interest and none in France.

Patient's typology (younger patient, no sequel, no disability) with Transient ischemic attack (TIA) and minor stroke (MS) makes them compatible with ambulatory management.

DETAILED DESCRIPTION:
Only two hospitals in France can take care patients with TIA or MS in an outpatient setting :Bichat hospital in Paris and Toulouse University Hospital. The effectiveness of this management has been demonstrated since recurrence stroke risk is reduced by 80% at one year. An English study (EXPRESS study) [2] showed a gain of 624 pounds with an ambulatory management compared to a conventional one. No studies are available in France on this subject.

The aim of this study is to test the feasibility of a collection of medical and economic data on a prospective way. The investigators collect medical (Cerebrovascular events, Stroke) and economic (direct and indirect costs) data concerning patients who were managed in TIA clinic in Toulouse Hospital. The medical data will be compiled with available French and International literature. The economic data will be compiled with available data in PMSI and health insurance database. This study aims to prepare a multicenter cohort to compare the cost effectiveness ratio between ambulatory and conventional management.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the TIA clinic in Toulouse Hospital (a day clinic)
* Having presented within the previous 7 days a transient ischemic attack or a minor stroke
* Affiliated to a social protection system
* To have given no opposition to participation in the study

Exclusion Criteria:

* Patients with a transient ischemic attack - mimic (such as migraine or seizure)
* Patients under protection of justice
* Pregnant and / or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients, to adapt to the recent change in the typology of new ischemic stroke in Western Europe, which for the most part are transient (30%) or minor ischemic strokes (35%). %).
  The profile of these patients is indeed compatible with outpatient care which should lead to the adaptation of the offer of care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The average cost-effectiveness ratio at 3 month | 3 months
  The average cost-effectiveness ratio at 3 month where the effectiveness is the 3-month cerebro vascular event rate and the costs taken into account are medical and non-medical direct costs and indirect costs limited to work stoppages.

SECONDARY OUTCOMES:
Percentage of full cost collection | 1 year
  Percentage of patients for whom total direct medical, direct non-medical, and indirect costs could be collected by comparing with health insurance data
Concordance between monitoring data collected in different database | 1 year
  Concordance between prospectively collected monitoring data, supplemented by data from the PMSI database of Toulouse University Hospital and data extracted from the health insurance database via NIR.
Recurrence rate of cerebro and cardiovascular events at 7 days | 7 days
  Recurrence rate of cerebro and cardiovascular events at 7 days : Stroke, myocardial infarction, vascular death within 30 days of stroke or MI
Recurrence rate of cerebro and cardiovascular events at 3 months | 3 months
  Recurrence rate of cerebro and cardiovascular events at 3 months : Stroke, myocardial infarction, vascular death within 30 days of stroke or MI
Recurrence rate of cerebro and cardiovascular events at one year | one year
  Recurrence rate of cerebro and cardiovascular events at one year : Stroke, myocardial infarction, vascular death within 30 days of stroke or MI
Average cost-effectiveness ratio at one year | one year
  The average cost - effectiveness ratio with the criterion of effectiveness the recurrence rate for cardiovascular events at one year (stroke, myocardial infarction, vascular death occurring within 30 days after a stroke or an IDM), and as cost criteria, direct medical and non-medical costs and indirect costs limited to work stoppages
Percentage of patients treated in TIA clinic who had first medical contact with a senior | 1 day
  Percentage of patients attending the AIT Clinic who had first medical contact with a senior neurology
Percentage of patients with statin prescription at discharge | 1 day
  Percentage of patients with statin prescription at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Derumeaux-Burel, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No